CLINICAL TRIAL: NCT03702582
Title: Trial of New Oral Anticoagulants vs. Warfarin for Post Cardiac Surgery Atrial Fibrillation
Brief Title: Rivaroxaban vs. Warfarin for Post Cardiac Surgery Atrial Fibrillation
Acronym: NEW-AF
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Asishana A Osho, Clinical Fellow in Surgery, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2018P002307
Record Dates: First submitted 2018-10-05; First posted 2018-10-11 (Actual); Last update posted 2023-10-24 (Actual); Status verified 2023-10

CONDITIONS: Atrial Fibrillation; Stroke; Bleeding
Keywords: Atrial Fibrillation; Rivaroxaban; Warfarin; Stroke; Anticoagulation; Bleeding
MeSH Terms: conditions — Atrial Fibrillation; Stroke; Hemorrhage | interventions — Rivaroxaban; Warfarin

STUDY DESIGN:
Intervention Model Description: Cardiac surgery patients who meet study criteria and develop recurrent or persistent atrial fibrillation post-operatively will be randomized 1:1 to receive Warfarin or Rivaroxaban for prophylaxis against stroke or other systemic arterial embolism
Masking Description: Statisticians performing comparative analyses of primary outcomes will be blinded as to the allocation designations of patients. Otherwise there will be no masking in the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Rivaroxaban (Experimental): Rivaroxaban: Direct inhibitor of Factor Xa, an enzyme that stimulates the formation of thrombin from prothrombin (A critical step in both the intrinsic and extrinsic aspects of the coagulation cascade)
  Dosage form: Per Os (Oral)
  Dosage and Frequency: 20 mg every evening with the evening meal (No titration requirements). For patients with decreased glomerular filtration rate (GFR between 15 ml/min and 50 ml/min), dosing will be decreased to 15 mg every evening with the evening meal.
  Duration: 30 days (Possibility of continuation after post-operative cardiology clinic visit)
  Interventions: Drug: Rivaroxaban
- Warfarin (Active Comparator): Warfarin: Competitive inhibitor of vitamin K epoxide reductase complex 1, an important enzyme in the activation pathway for vitamin K dependent coagulation factors
  Dosage form: Per Os (Oral)
  Dosage and Frequency: Initial dose of 2 - 5 mg nightly after the evening meal (QHS) with appropriate titration to goal INR 2.0 - 3.0 (Initial dose based on weight, age, gender, co-morbidities and concurrent medications). INR will be checked daily to weekly depending on stability of dosing and medication regimen.
  Duration: 30 days (Possibility of continuation after post-operative Cardiology clinic visit)
  Interventions: Drug: Warfarin

INTERVENTIONS:
Drug: Rivaroxaban — Anticoagulant drug that works via direct inhibition of factor Xa. FDA approved for prophylaxis against stroke in non-valvular atrial fibrillation
  Other Names: Xarelto; Database of Molecules (PubChem CID): 6433119
  Arms: Rivaroxaban
Drug: Warfarin — Anticoagulation drug that works via inhibition of vitamin K dependent clotting factors. FDA approved for prophylaxis against stroke in atrial fibrillation
  Other Names: Coumadin; Database of Molecules (PubChem CID): 54678486
  Arms: Warfarin

SUMMARY:
This prospective, randomized, active-controlled, parallel arm study compares the safety and financial benefits of arterial thromboembolism prophylaxis with Warfarin vs. Rivaroxaban (A novel oral anticoagulant) in patients with new onset atrial fibrillation after sternotomy for cardiac operations.

DETAILED DESCRIPTION:
New onset atrial fibrillation (NOAF) is a common occurrence following cardiac surgery, occurring in 20-30% of patients post-operatively. Historically, Vitamin K antagonist therapy with Warfarin has been the treatment of choice for prophylaxis against stroke and systemic arterial thromboembolism in NOAF. Warfarin inhibits the Vitamin K dependent factors involved in both the intrinsic and extrinsic coagulation cascades, thus decreasing systemic clotting. However, Warfarin therapy comes with many challenges including prolonged titration, tedious monitoring requirements and in some cases, increased bleeding risk.

The limitations associated with Warfarin may be mitigated by using new oral anticoagulants (NOACs) like Rivaroxaban which have no routine monitoring requirements. Rivaroxaban is a direct inhibitor of Factor Xa, a central reactant in both the intrinsic and extrinsic coagulation cascades. Studies in non-operative patients with atrial fibrillation have shown that Rivaroxaban is non-inferior to Warfarin for stroke prophylaxis with similar risk profiles. This study aims to compare the efficacy, safety and financial cost of these two drugs when used for the management of new onset atrial fibrillation that occurs after cardiac operations.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female ≥ 18 years
* At least one of the following procedures: coronary artery bypass grafting, aortic valve repair, mitral valve repair, non-mechanical aortic valve replacement, any combination of these procedures
* Two or more episodes of New Onset Atrial Fibrillation (each lasting > 20 minutes) or persistent atrial fibrillation lasting > 24 hours (Or for >18 hours over a 24-hour interval)
* If female of child-bearing age, use of adequate contraception

Exclusion Criteria:

* Pre-existing paroxysmal atrial fibrillation before cardiac surgery
* Pre-existing indications for therapeutic anticoagulation (Including but not limited to PE, DVT, mechanical valve)
* Moderate-to-severe mitral valve stenosis not surgically corrected
* Pre-existing allergy to study medications
* Recent (< 1 year) or ongoing pregnancy (Urine pregnancy test will be obtained for women of child bearing age at the time of enrollment into the study)
* Stroke within 1 month prior to surgery or postoperatively prior to initiation of study drugs
* Postoperative bleeding episode prior to initiation of study drug
* Severe dysfunction of another organ system including GFR < 30 ml/min, baseline INR > 1.7, ileus or other gastrointestinal pathology hindering ability to absorb oral medications, and known coagulation pathway deficiencies
* Postoperative need for non-aspirin anti-platelet therapy that cannot be discontinued when therapeutic anticoagulation is initiated
* Patient taking medications with known major interactions with study drugs with no therapeutic alternatives)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2019-04-30 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2023-10-01 (Actual)

PRIMARY OUTCOMES:
Postoperative Length of Stay | Up to 6 months following the cardiac operation
  Length of inpatient stay in days from time of departure from the operating room

SECONDARY OUTCOMES:
Episode of Major Bleeding (Defined as the occurrence of any of several events listed in the description. No specific scale, questionnaire or instrument will be used) | Up to 30 days after discharge from the initial postoperative hospitalization
  Major bleeding defined as re-operation or other therapeutic intervention for bleeding (including but not limited to colonoscopy, upper endoscopy and urologic procedures for hematuria), development of any intracranial bleeding, cessation of study drug for bleeding concerns, reversal of study drug for bleeding concerns and/or new transfusion requirement > 2 units of blood after drug administration
Cerebrovascular accident (CVA) | Up to 30 days after discharge from the initial postoperative hospitalization
  Rates of cerebrovascular accident including stroke and transient ischemic attack (TIA)
Other systemic embolism | Up to 30 days after discharge from the initial postoperative hospitalization
  Rates of non-neurological systemic arterial embolism involving any organ system
Deep venous thrombosis (DVT) and/or Pulmonary Embolism (PE) | Up to 30 days after discharge from the initial postoperative hospitalization
  Occurrence of pathologic venous thrombo-embolism including DVT and PE
Minor Bleeding | Up to 30 days after discharge from the initial postoperative hospitalization
  Minor bleeding defined as blood transfusions <= 2 units or drop in hemoglobin greater 3g/dL following administration of study drugs
Number of Transfusions | Up to 30 days after discharge from the initial postoperative hospitalization
  The number of units of blood transfused for each participant after initiation of study drugs
Hospital Readmission | Up to 30 days after discharge from the initial postoperative hospitalization
  Readmissions will be counted in this calculation if patients are admitted to the hospital. Emergency room visits without admission and outpatient visits will not count toward this calculation of readmission rates.
Therapy related costs of anticoagulation | Up to 30 days after discharge from the initial postoperative hospitalization
  Specific drug related costs will be estimated in dollars for patients in each intervention arm. This will include costs of all administered drug doses as well as costs of associated laboratory studies and mileage based costs of travel to INR testing centers
Performance on the EUROQOL (EQ-5D) Quality of Life Instrument | Up to 30 days after discharge from the initial postoperative hospitalization
  Participants will be administered the EUROQOL-5D-3L (5 dimensions, 3 levels) questionnaire to derive an estimate of the health state. This is comprised of a 5 questions survey and a single visual analog scale highlighting perceived health levels
  For the 5 questions survey, each question related to mobility, selfcare, mood, pain and/or functionality is answered on a three point scale with higher number representing worse outcomes. The entire dataset is used to generate a health state based on the unique pattern of answers. These health states are then compared against standardized country-based value sets which provide an assessment of quality of life based on societal preferences.
  The visual analog scale is single answer between 0 and 100 representing the patient's perception of their health state. 0 represents the worst health imaginable and 100 represents the best.
Average score on the Perception of Anticoagulant Treatment Questionnaire (PACT-Q2) | Up to 30 days after discharge from the initial postoperative hospitalization
  Participants will be administered the PACT-Q2 questionnaire which is comprised of a convenience subscale and a satisfaction subscale.
  For the convenience subscale, each of 13 questions is answered on a 1-5 rating scale with higher numbers representing worse outcomes. A sub-scale score is generated by inverting the score from each element and calculating the sum. Range on the inverted scale is 13 - 65. Higher scores represent better outcomes.
  For the satisfaction subscale, each of 7 questions is answered on a 1-5 rating scale with higher numbers representing better outcomes. The total score on this subscale is generated by adding up scores from all elements. Range on this subscale is 7-35. Higher scores represent better outcomes.
  A composite score is generated by adding up scores from both subscales and recalibrating on a 0-100 scale by adding the scores together and applying the formula: COMPOSITE SCORE=100×(Sum-20)/80. Higher scores represent more favorable outcomes.
Rate of ongoing atrial fibrillation | Up to 30 days after discharge from the initial postoperative hospitalization
  EKGs will be obtained at various time points during the study to determine whether participants remain in atrial fibrillation during the follow up period. From each EKG, existence of p-waves, regularity of the overall wave form and heart rate will be evaluated to determine if patients remain in atrial fibrillation or if they have spontaneously converted to a normal sinus rhythm.
Rate of Mortality | Up to 30 days after discharge from the initial postoperative hospitalization
  Mortality during study follow up will be documented and rates will compared across intervention groups. Cause of death will be documented
Rates of adverse clinical outcomes | Up to 30 days after discharge from the initial postoperative hospitalization
  Other adverse clinical outcomes will be documented and rates compared between intervention arms including: Acute Kidney Injury, Infection, Heart Failure, Pericardial Effusion, Myocardial infarction, Pleural Effusion and Hepatic dysfunction

CONTACTS AND LOCATIONS:
Overall Officials: Asishana A Osho, MD, MPH, Principal Investigator — Massachusetts General Hospital; Thoralf M Sundt, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided
At this time there is no plan to make Individual Participant Data available to other researchers. As the study develops, investigators will consider making an individual participant data sharing plan if there is interest from other researchers.

REFERENCES:
- [Background] Spyropoulos AC, Ageno W, Albers GW, Elliott CG, Halperin JL, Hiatt WR, Maynard GA, Steg PG, Weitz JI, Suh E, Spiro TE, Barnathan ES, Raskob GE; MARINER Investigators. Rivaroxaban for Thromboprophylaxis after Hospitalization for Medical Illness. N Engl J Med. 2018 Sep 20;379(12):1118-1127. doi: 10.1056/NEJMoa1805090. Epub 2018 Aug 26. PMID 30145946
- [Background] Butt JH, Xian Y, Peterson ED, Olsen PS, Rorth R, Gundlund A, Olesen JB, Gislason GH, Torp-Pedersen C, Kober L, Fosbol EL. Long-term Thromboembolic Risk in Patients With Postoperative Atrial Fibrillation After Coronary Artery Bypass Graft Surgery and Patients With Nonvalvular Atrial Fibrillation. JAMA Cardiol. 2018 May 1;3(5):417-424. doi: 10.1001/jamacardio.2018.0405. PMID 29590304
- [Background] Charlton B, Adeboyeje G, Barron JJ, Grady D, Shin J, Redberg RF. Length of hospitalization and mortality for bleeding during treatment with warfarin, dabigatran, or rivaroxaban. PLoS One. 2018 Mar 28;13(3):e0193912. doi: 10.1371/journal.pone.0193912. eCollection 2018. PMID 29590141
- [Background] Megens MR, Churilov L, Thijs V. New-Onset Atrial Fibrillation After Coronary Artery Bypass Graft and Long-Term Risk of Stroke: A Meta-Analysis. J Am Heart Assoc. 2017 Dec 22;6(12):e007558. doi: 10.1161/JAHA.117.007558. PMID 29273637
- [Background] Hawks MK, Bryce C. Rivaroxaban vs. Warfarin for Anticoagulation in Patients with Atrial Fibrillation Undergoing Ablation and Cardioversion. Am Fam Physician. 2016 Oct 1;94(7):Online. No abstract available. PMID 27929207
- [Background] Gillinov AM, Bagiella E, Moskowitz AJ, Raiten JM, Groh MA, Bowdish ME, Ailawadi G, Kirkwood KA, Perrault LP, Parides MK, Smith RL 2nd, Kern JA, Dussault G, Hackmann AE, Jeffries NO, Miller MA, Taddei-Peters WC, Rose EA, Weisel RD, Williams DL, Mangusan RF, Argenziano M, Moquete EG, O'Sullivan KL, Pellerin M, Shah KJ, Gammie JS, Mayer ML, Voisine P, Gelijns AC, O'Gara PT, Mack MJ; CTSN. Rate Control versus Rhythm Control for Atrial Fibrillation after Cardiac Surgery. N Engl J Med. 2016 May 19;374(20):1911-21. doi: 10.1056/NEJMoa1602002. Epub 2016 Apr 4. PMID 27043047
- [Background] Anderson E, Johnke K, Leedahl D, Glogoza M, Newman R, Dyke C. Novel oral anticoagulants vs warfarin for the management of postoperative atrial fibrillation: clinical outcomes and cost analysis. Am J Surg. 2015 Dec;210(6):1095-102; discussion 1102-3. doi: 10.1016/j.amjsurg.2015.07.005. Epub 2015 Sep 18. PMID 26482512
- [Background] Giugliano RP, Ruff CT, Braunwald E, Murphy SA, Wiviott SD, Halperin JL, Waldo AL, Ezekowitz MD, Weitz JI, Spinar J, Ruzyllo W, Ruda M, Koretsune Y, Betcher J, Shi M, Grip LT, Patel SP, Patel I, Hanyok JJ, Mercuri M, Antman EM; ENGAGE AF-TIMI 48 Investigators. Edoxaban versus warfarin in patients with atrial fibrillation. N Engl J Med. 2013 Nov 28;369(22):2093-104. doi: 10.1056/NEJMoa1310907. Epub 2013 Nov 19. PMID 24251359
- [Background] Granger CB, Alexander JH, McMurray JJ, Lopes RD, Hylek EM, Hanna M, Al-Khalidi HR, Ansell J, Atar D, Avezum A, Bahit MC, Diaz R, Easton JD, Ezekowitz JA, Flaker G, Garcia D, Geraldes M, Gersh BJ, Golitsyn S, Goto S, Hermosillo AG, Hohnloser SH, Horowitz J, Mohan P, Jansky P, Lewis BS, Lopez-Sendon JL, Pais P, Parkhomenko A, Verheugt FW, Zhu J, Wallentin L; ARISTOTLE Committees and Investigators. Apixaban versus warfarin in patients with atrial fibrillation. N Engl J Med. 2011 Sep 15;365(11):981-92. doi: 10.1056/NEJMoa1107039. Epub 2011 Aug 27. PMID 21870978
- [Background] Patel MR, Mahaffey KW, Garg J, Pan G, Singer DE, Hacke W, Breithardt G, Halperin JL, Hankey GJ, Piccini JP, Becker RC, Nessel CC, Paolini JF, Berkowitz SD, Fox KA, Califf RM; ROCKET AF Investigators. Rivaroxaban versus warfarin in nonvalvular atrial fibrillation. N Engl J Med. 2011 Sep 8;365(10):883-91. doi: 10.1056/NEJMoa1009638. Epub 2011 Aug 10. PMID 21830957
- [Background] Connolly SJ, Ezekowitz MD, Yusuf S, Eikelboom J, Oldgren J, Parekh A, Pogue J, Reilly PA, Themeles E, Varrone J, Wang S, Alings M, Xavier D, Zhu J, Diaz R, Lewis BS, Darius H, Diener HC, Joyner CD, Wallentin L; RE-LY Steering Committee and Investigators. Dabigatran versus warfarin in patients with atrial fibrillation. N Engl J Med. 2009 Sep 17;361(12):1139-51. doi: 10.1056/NEJMoa0905561. Epub 2009 Aug 30. PMID 19717844
- [Derived] Osho AA, Moonsamy P, Ethridge BR, Leya GA, D'Alessandro DA, Jassar AS, Villavicencio MA, Melnitchouk SI, Tolis G, Langer NB, Funamoto M, Li SS, Colon KM, Mohan N, Locascio JJ, Lubitz SA, Akeju O, Sundt TM. Rationale and Design of the Randomized Controlled Trial of New Oral Anticoagulants Versus Warfarin for Post Cardiac Surgery Atrial Fibrillation: The NEW-AF Trial. Ann Surg. 2022 Jul 1;276(1):200-204. doi: 10.1097/SLA.0000000000004459. Epub 2020 Sep 1. PMID 32889881